CLINICAL TRIAL: NCT03411954
Title: Hippocampus Avoidance During Intensity Modulated Radiotherapy for T4 Nasopharyngeal Carcinoma Patients:an Open, Prospective,Non-randomized Phase III Clinical Trial
Brief Title: Hippocampus Avoidance During Intensity Modulated Radiotherapy for T4 Nasopharyngeal Carcinoma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NPC-2017-209
Record Dates: First submitted 2018-01-13; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: hippocampus avoidance; cognitive changes; intensity modulated radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HP-RT: Hippocampus avoidance: decrease the dose to hippocampus as low as possible without affecting the target volumes and other normal tissues

SUMMARY:
This is a prospective, non-randomized phase III study observing the cognitive function changes with conformal hippocampus avoidance during intensity modulated radiotherapy for T4 nasopharyngeal carcinoma patients.

DETAILED DESCRIPTION:
All patients received intensity modulated radiotherapy or Tomotherapy with or without chemotherapy. Before radiotherapy, the patients will receive brain MRI scanning and the brain MRI images will be fused with the head and neck CT scan images. The investigators develop the treatment plan with hippocampus avoidance. Cognitive function are evaluated before,during and after radiotherapy. Dose-volume Histograms are got to analyze the associated factors.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologic confirmed nasopharyngeal carcinoma
2. ECOG performance scale 0-2
3. Tumor stage is T4N0-3M0-1 according to 8th American Joint Commission on Cancer edition
4. Adequate hepatic, renal and hematologic functions (hemoglobin ≥ 90g/L, platelets ≥ 100×10^9/L, neutrophils ≥ 1.5×10^9/L, serum transaminase < 2.5×the upper limit of normal(ULN), (If liver metastases, serum transaminase< 5×the ULN), creatinine clearance rate > 60ml/min.
5. Informed consent signed.

Exclusion Criteria:

1. History of malignant tumors.
2. Any severe complications contraindicated chemotherapy or radiotherapy.
3. Medical history of central nervous system, cognitive or psychological diseases;
4. Pregnant or nursing women.
5. Patients with mental disease cannot complete the questionaire.
6. MRI contraindication -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
the dose-volume relationship between hippocampus and cognitive function | 1 year
  To explore the relationship between cognitive impairment and exposure dose of hippocampus in patients with nasopharyngeal carcinoma.

SECONDARY OUTCOMES:
cognitive function changes | 1 year
  response to the Montreal Cognitive Assessment
memory function changes | 1 year
  response to the Hopkins Verbal Learning Test
quality of life | 1 year
  response to the QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: yuanyaun chen, professor, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No